CLINICAL TRIAL: NCT05906264
Title: Evaluation of Compliance and Effectiveness of Pulmonary Rehabilitation Program in COPD Patient
Brief Title: Pulmonary Rehabilitation Program in COPD Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC_COPD_Rehab
Record Dates: First submitted 2022-04-19; First posted 2023-06-15 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation; Tele-rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Compared to control group, interventional group will be provided tele-intervention every week, checking compliance and encouraging the rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulmonary rehabilitation, Control (No Intervention): for COPD patients, who have been trained with the pulmonary rehabilitation program
  * Compliance will be checked by monitoring wearable device at one month
  * Pulmonary function and symptom improvement effect will be checked at 3 months
- Pulmonary rehabilitation, Intervention (Active Comparator): Compared to Control group, Intervention group will be provided with additional tele-intervention every week to check the compliance and encourage of the rehabilitation
  Interventions: Behavioral: Tele-intervention

INTERVENTIONS:
Behavioral: Tele-intervention — Tele-intervention every week to check compliance and encourage the rehabilitation
  Arms: Pulmonary rehabilitation, Intervention

SUMMARY:
This study was designed in order to evaluate the compliance of a pulmonary rehabilitation program using a wearable device and the application effect of the program according to the characteristics of each patient, in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by persistent respiratory symptoms and airflow limitation. Symptoms of COPD often restricts exercise capacity and activities of daily life of patients. Accordingly, patients with symptomatic COPD have reduced health-related quality of life, which leads to substantial socioeconomic burden.

In order to overcome the limitation associated with COPD pharmacotherapy, the need for a combination of nonpharmacologic therapies, including pulmonary rehabilitation has been suggested constantly. Pulmonary rehabilitation is a method of relieving respiratory distress symptoms through exhalation and inspiratory training, improving exercise ability and contributes in improving lung function and overall quality of life.

Nevertheless, compliance of pulmonary rehabilitation in daily life is low in most COPD patients. Thus, we applied wearable device to detect and evaluate application, compliance and effectiveness pulmonary rehabilitation program in COPD patients, according to the patients' characteristics. Moreover, we sought to use the results of this study as a basic data to establish a strategy for a customized education program for each patient that can be applied to non-face-to-face digital therapeutics in the future.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients 18 years of age or older
* ECOG PS (Eastern Cooperative Oncology Group Performance Status) <2
* Smart phone user
* Those who understand the contents of the questionnaire and agree to the research

Exclusion Criteria:

* Patients with history of lung cancer surgery
* Patients with bronchiectasis, severe tuberculosis destroyed lung, active pulmonary tuberculosis, non-tuberculous mycobacterial lung disease (NTM), and idiopathic interstitial pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Activity minutes in 1 month | 1 month after training
  metabolic equivalents (METs)/day
Pulmonary function test | 1 month after training
  Maximum phonation time (seconds)
Dyspnea scale | 1 month after training
  mMRC dyspnea scale (0-4)

SECONDARY OUTCOMES:
Activity minutes in 3 months | 3 month after training
  metabolic equivalents (METs)/day
Pulmonary function test | 3 month after training
  Pulmonary function test (FEV1/FVC)
Dyspnea scale | 3 month after training
  mMRC dyspnea scale (0-4)
Functional capacity | 3 month after training
  6 minute walk test (m/6min)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Background] Mirza S, Clay RD, Koslow MA, Scanlon PD. COPD Guidelines: A Review of the 2018 GOLD Report. Mayo Clin Proc. 2018 Oct;93(10):1488-1502. doi: 10.1016/j.mayocp.2018.05.026. PMID 30286833
- [Background] Eisner MD, Anthonisen N, Coultas D, Kuenzli N, Perez-Padilla R, Postma D, Romieu I, Silverman EK, Balmes JR; Committee on Nonsmoking COPD, Environmental and Occupational Health Assembly. An official American Thoracic Society public policy statement: Novel risk factors and the global burden of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 Sep 1;182(5):693-718. doi: 10.1164/rccm.200811-1757ST. PMID 20802169
- [Background] Mathioudakis AG, Janssens W, Sivapalan P, Singanayagam A, Dransfield MT, Jensen JS, Vestbo J. Acute exacerbations of chronic obstructive pulmonary disease: in search of diagnostic biomarkers and treatable traits. Thorax. 2020 Jun;75(6):520-527. doi: 10.1136/thoraxjnl-2019-214484. Epub 2020 Mar 26. PMID 32217784
- [Background] Simmering JE, Polgreen LA, Comellas AP, Cavanaugh JE, Polgreen PM. Identifying Patients With COPD at High Risk of Readmission. Chronic Obstr Pulm Dis. 2016 Aug 29;3(4):729-738. doi: 10.15326/jcopdf.3.4.2016.0136. PMID 28848899
- [Background] Miravitlles M, Murio C, Guerrero T, Gisbert R; DAFNE Study Group. Decisiones sobre Antibioticoterapia y Farmacoeconomia en la EPOC. Pharmacoeconomic evaluation of acute exacerbations of chronic bronchitis and COPD. Chest. 2002 May;121(5):1449-55. doi: 10.1378/chest.121.5.1449. PMID 12006427
- [Background] Ko FW, Chan KP, Hui DS, Goddard JR, Shaw JG, Reid DW, Yang IA. Acute exacerbation of COPD. Respirology. 2016 Oct;21(7):1152-65. doi: 10.1111/resp.12780. Epub 2016 Mar 30. PMID 27028990
- [Background] Zeng Y, Jiang F, Chen Y, Chen P, Cai S. Exercise assessments and trainings of pulmonary rehabilitation in COPD: a literature review. Int J Chron Obstruct Pulmon Dis. 2018 Jun 26;13:2013-2023. doi: 10.2147/COPD.S167098. eCollection 2018. PMID 29983556
- [Background] Lacasse Y, Goldstein R, Lasserson TJ, Martin S. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD003793. doi: 10.1002/14651858.CD003793.pub2. PMID 17054186
- [Background] Ribeiro F, Theriault ME, Debigare R, Maltais F. Should all patients with COPD be exercise trained? J Appl Physiol (1985). 2013 May;114(9):1300-8. doi: 10.1152/japplphysiol.01124.2012. Epub 2013 Feb 14. PMID 23412902
- [Background] Oga T, Nishimura K, Tsukino M, Hajiro T, Mishima M. Dyspnoea with activities of daily living versus peak dyspnoea during exercise in male patients with COPD. Respir Med. 2006 Jun;100(6):965-71. doi: 10.1016/j.rmed.2005.10.006. Epub 2005 Nov 18. PMID 16298519
- [Background] Bianchi R, Gigliotti F, Romagnoli I, Lanini B, Castellani C, Binazzi B, Stendardi L, Bruni GI, Scano G. Impact of a rehabilitation program on dyspnea intensity and quality in patients with chronic obstructive pulmonary disease. Respiration. 2011;81(3):186-95. doi: 10.1159/000273675. Epub 2010 Jan 5. PMID 20090282
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694